CLINICAL TRIAL: NCT01725815
Title: A Peer-Led, Medical Disease Self-Management Program for Mental Health Consumers
Brief Title: The Health Access and Recovery Peer Program
Acronym: HARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Druss, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00047631a; 1R01MH090584-01A1 (NIH)
Record Dates: First submitted 2012-04-25; First posted 2012-11-14 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Hypertension; Arthritis; Coronary Artery Disease; Hepatitis; Diabetes; Asthma; Hyperlipidemia; HIV
MeSH Terms: conditions — Hypertension; Arthritis; Coronary Artery Disease; Hepatitis; Diabetes Mellitus; Asthma; Hyperlipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HARP Intervention (Experimental)
  Interventions: Behavioral: HARP Intervention
- No Intervention: Control (No Intervention): Participants in usual care will continue to obtain any mental health or peer-support services that they would otherwise be receiving.

INTERVENTIONS:
Behavioral: HARP Intervention — The HARP intervention is a 6-week, 6-session, group format intervention to improve self-management of chronic medical diseases. Each group lasts 90 minutes and has 8-12 attendees. Between groups, participants work with partners from the group to troubleshoot problems and accomplish action plans identified during the session. At the end of the program, monthly alumni groups meet for six months to reinforce lessons from the intervention, monitor progress, and maintain peer support.
  Arms: HARP Intervention

SUMMARY:
Individuals with serious mental illnesses (SMI) face high rates of medical comorbidity as well as challenges in managing these conditions. A growing workforce of certified peer specialists is available to help these individuals more effectively manage their health and health care. However, there is little existing research examining the effectiveness of peer-led medical self-management programs for this population. in this trial, participants were randomized to either the Health and Recovery Peer program (HARP), a medical disease self-management program led by certified peer specialists, or to care as usual. Assessments were conducted at baseline, 3 months, and 6 months.

DETAILED DESCRIPTION:
Persons with serious mental illnesses (SMI) face elevated rates of medical comorbidity, and also challenges in effectively managing these health problems. There is an urgent need to develop self-management strategies that allow persons with SMI to more effectively manage their chronic medical illnesses.

In general populations, peer-led disease self-management interventions have been demonstrated to be feasible, effective, scalable, and to lead to sustainable improvements in self-management and health outcomes. With funding from an R34 intervention development grant from NIMH, the study team has developed and piloted a modified version of the most widely tested and used peer-led self management program, the Chronic Disease Self-Management Program (CDSMP), for persons with serious mental illness. Two pilot tests of this intervention, the Health and Recovery Peer (HARP) program, demonstrated that the program can be implemented with high engagement, retention, and program fidelity, and can result in effect sizes across a range of outcomes comparable to or greater than those seen in general medical populations.

This application proposes to conduct a fully-powered, multisite trial of the HARP program. A total of 400 individuals with serious mental illnesses and one or more chronic medical condition will be recruited from three diverse community mental health clinics in the Atlanta metro region and randomized to the HARP program or usual care. For individuals in the HARP program, two peer educators with SMI and one or more chronic medical condition will lead a six-session, six-week manualized intervention, which helps participants become more effective managers of their chronic illnesses. Follow-up interviews and chart reviews at 3 months, 6 months and one year will assess changes in clinical outcomes, improvement in generic and disease-specific measures of illness self-management, and quality of care. During the final phase of the study, a dissemination strategy building on the CDSMP training infrastructure will allow program participants to lead HARP groups.

This study will establish the first fully peer-led, evidence-based intervention for improving physical self-management in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* On CMHC roster of active patients.
* Presence of a serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder, major depression, obsessive-compulsive disorder, or post-traumatic stress disorder
* Chronic Medical Condition as noted in the CMHC chart or via self-report: (hypertension; arthritis; heart disease; diabetes; and asthma/COPD),

Exclusion Criteria:

* cognitive impairment based on a score of > 3 on a 6-item, validated screener developed for clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06-01 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Druss, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Central Fulton Community Mental Health Center at Grady Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HARP Intervention | No Intervention: Control
Started | 198 | 202
Completed | 198 | 202
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HARP Intervention | No Intervention: Control | Total
Number analyzed (Participants) | 198 | 202 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.74 (8.72) | 49.69 (9.51) | 49.71 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 123 | 255
  Male | 66 | 79 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 131 | 133 | 264
  White | 60 | 60 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 198 | 202 | 400
Total annual Income [Count of Participants; unit: Participants]
  $0-$5000 | 96 | 87 | 183
  $5000-$10000 | 53 | 60 | 113
  $10000-$15000 | 26 | 27 | 53
  >$15000 | 21 | 24 | 45
  Unknown | 2 | 4 | 6
Insurance status [Count of Participants; unit: Participants]
  Medicaid | 56 | 60 | 116
  Medicare | 38 | 47 | 85
  Private insurance | 6 | 14 | 20
  Unknown | 98 | 81 | 179
Medical Diagnosis [Count of Participants; unit: Participants]
  Diabetes | 51 | 65 | 116
  Heart Disease/CAD/CHD | 25 | 20 | 45
  Hyperlipidemia | 81 | 82 | 163
  Hypertension | 133 | 142 | 275
  Arthritis | 93 | 79 | 172
  Hepatitis | 19 | 25 | 44
  Asthma/COPD | 65 | 72 | 137
  HIV | 6 | 12 | 18
Primary Mental Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia/Schizoaffective | 52 | 62 | 114
  Bipolar Disorder | 74 | 80 | 154
  Depression | 141 | 139 | 280
  Obsessive Compulsive Disorder | 12 | 18 | 30
  Post-Traumatic stress Disorder | 43 | 58 | 101

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life (HRQOL)
Description: The short form-36-item (SF-36) Physical component score (PCS) is a measure of HRQOL constructed for use in the Medical Outcomes Study that rely upon patient self-reporting and reflects the physical functioning. The scores ranges from 0-100 with higher scores indicating greater levels of physical functioning.
Time Frame: Baseline, 3 months post-intervention, 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARP Intervention | No Intervention: Control
Number analyzed (Participants) | 198 | 202
score on a scale
  Baseline | 32.73 (10.92) | 32.74 (11.29)
  3 months post-intervention | 34.49 (11.15) | 33.89 (10.41)
  6 months post-intervention | 35.42 (11.02) | 34.15 (11.52)

2. Secondary Outcome: Behavioral Activation
Description: Behavioral Activation was measured using the Patient Activation Measure (PAM), an instrument which has been found to be reliable and valid across a wide range of patient populations. The Patient Activation Measure (PAM) is a 22-item measure that assesses patient knowledge, skill, and confidence for self-management. Possible scores range from 0 to 100, with higher scores indicating greater patient activation (better outcome).
Time Frame: Baseline, 3 months post-intervention, 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARP Intervention | No Intervention: Control
Number analyzed (Participants) | 198 | 202
score on a scale
  Baseline | 57.4 (16.6) | 55.7 (14.9)
  3 months post-intervention | 61.6 (15.9) | 56.4 (16.5)
  6 months post-intervention | 60.5 (16.7) | 57.2 (16.3)

3. Secondary Outcome: Dietary Intake
Description: Dietary intake was assessed with the Block Fat-Sugar-Fruit-Vegetable Screener, which is a validated 55-item scale assessing both frequency and quantity of food intake based on typical eating habits. Possible scores range from 0 to 68, with higher scores indicating greater consumption of fat (worse outcome).
Time Frame: Baseline, 3 months post-intervention, 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARP Intervention | No Intervention: Control
Number analyzed (Participants) | 198 | 202
score on a scale
  Baseline | 10.1 (5.1) | 9.8 (5.6)
  3 months post-intervention | 10.1 (5.0) | 9.3 (5.3)
  6 months post-intervention | 10.2 (5.6) | 9.4 (5.3)

4. Secondary Outcome: Medication Adherence
Description: Medication Adherence was assessed using the Morisky scale, a 4-item questionnaire that has been shown to have strong content and predictive validity in hypertension,cardiovascular disease,and diabetes. Possible scores range from 0 to 4 with lower scores indicating greater medication adherence.
Time Frame: Baseline, 3 months post-intervention, 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARP Intervention | No Intervention: Control
Number analyzed (Participants) | 198 | 202
score on a scale
  Baseline | 0.92 (0.94) | 0.94 (1.02)
  3 months post-intervention | 0.79 (0.92) | 0.97 (0.96)
  6 months post-intervention | 0.84 (0.92) | 0.89 (0.96)

ADVERSE EVENTS:
Time Frame: 3 months post-intervention, 6 months post-intervention
Arm/Group | HARP Intervention | No Intervention: Control
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/202
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/202
Other Adverse Events (participants affected / at risk) | 0/198 | 0/202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT01725815/Prot_SAP_000.pdf